CLINICAL TRIAL: NCT04100512
Title: Oscillating Positive Expiratory Pressure (OPEP) Therapy in Trauma Patients With Multiple Rib Fractures: A Randomized Comparative Trial Against Incentive Spirometry
Brief Title: Oscillating Positive Expiratory Pressure (OPEP) Therapy in Trauma Patients With Multiple Rib Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poudre Valley Health System (Other)
Collaborators: Monaghan Medical Corporation (Unknown)
Responsible Party: Principal Investigator, Julie Dunn, M.D., Trauma Research Medical Director, Poudre Valley Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPEP7292019
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Rib Fractures; Respiratory Complication
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Incentive spirometry (Active Comparator): Each patient will be instructed on how to use the respiratory therapy device, either IS or OPEP, by research personnel and respiratory therapists. Participants will be instructed to record their compliance with the RT protocol in their respective patient diaries. Patient diaries will be collected upon discharge for analysis.
  Interventions: Device: Incentive spirometry
- Oscillating Positive Expiratory Pressure Device (Experimental): Each patient will be instructed on how to use the respiratory therapy device, either IS or OPEP, by research personnel and respiratory therapists. Participants will be instructed to record their compliance with the RT protocol in their respective patient diaries. Patient diaries will be collected upon discharge for analysis.
  Interventions: Device: Oscillating Positive Expiratory Pressure Device

INTERVENTIONS:
Device: Oscillating Positive Expiratory Pressure Device — Aerobika® Oscillating Positive Expiratory Pressure (OPEP) device is a drug-free, easy to use, hand-held device with a proprietary pressure-oscillation dynamic that provides intermittent resistance and creates positive pressure and oscillations simultaneously. The Aerobika® OPEP device opens weak or collapsed airways to mobilize and assist mucociliary clearance to the upper airways where it can be coughed out.
  Arms: Oscillating Positive Expiratory Pressure Device
Device: Incentive spirometry — An incentive spirometer is a device that measures how deeply you can inhale (breathe in). It helps you take slow, deep breaths to expand and fill your lungs with air. The incentive spirometer is made up of a breathing tube, an air chamber, and an indicator.
  Arms: Incentive spirometry

SUMMARY:
To determine the efficacy of oscillatory positive expiratory pressure (OPEP) therapy on patients admitted through the trauma service line for rib fractures, as compared to incentive spirometry (IS).

DETAILED DESCRIPTION:
Patients identified through screening procedures to fit the inclusion criteria will be approached, within 48 hours of floor admission, to participate in the study. Once written informed consent is obtained, participants will be randomized, in a 1:1 ratio, into either the IS or OPEP study group.

Each patient will be instructed on how to use the respiratory therapy device, either IS or OPEP, by research personnel and respiratory therapists. Participants will be instructed to record their compliance with the RT protocol in their respective patient diaries.

Respiratory Therapy will record FVC three times daily on all study participants until stable (FVC > 1.5L x 4), then daily for up to 7 days or until discharge.

Participants will be contacted on day 30 from discharge, and administered a short questionnaire. All participants will be followed and monitored per standard of care, under the care and supervision of their treating provider teams.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Greater than or equal to 1 Rib Fracture
* Admitted to trauma services at Medical Center of the Rockies (MCR).

Exclusion Criteria:

* Less than 18 years old
* Any physical injury that creates inability to functionally use devices
* Adults unable to consent or cooperate due to
* Dementia
* Confusion
* On ventilator support
* Moderate to severe Traumatic brain injury (Glasgow Coma Scale < 12)
* Cervical spinal cord injury
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Time (hours) to stable forced vital capacity | 3 times daily, until FVC is >1.5 liters x 4 consecutive tests, or up to 4 weeks
  Time (hours) to stable forced vital capacity (FVC) defined as >1.5 liters x 4 tests and FVC at 7 days for both IS and OPEP participants.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dunn, MD, Principal Investigator — Trauma Research Medical Director
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States